CLINICAL TRIAL: NCT06445699
Title: Investigation the Clinical Effectiveness of Combination Topical Aminolaevulinic Acid-Photodynamic Therapy With Hydrogel Dressing for Treatment Chronic Cutaneous Wounds
Brief Title: Photodynamic Therapy With Hydrogel Dressing for Chronic Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Rui Yin, MD, PhD, Army Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYin
Record Dates: First submitted 2024-05-21; First posted 2024-06-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Photodynamic Therapy
Keywords: Wound healing; Aminolaevulinic acid; Photodynamic therapy; Hydrogel dressing
MeSH Terms: interventions — Photochemotherapy; Bandages, Hydrocolloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Grp.1) (Active Comparator): The patients received hydrogel dressing change at three days intervals
  Interventions: Other: Hydrogel dressing
- Group 2 (Grp.2) (Experimental): The patients received ALA-PDT treatment at ten days intervals for 4 sessions.
  Interventions: Other: Photodynamic therapy
- Group 3 (Grp.3) (Experimental): The patients received ALA-PDT at ten days intervals for 4 sessions combined with hydrogel dressing change every three days intervals.
  Interventions: Other: Photodynamic therapy; Other: Hydrogel dressing

INTERVENTIONS:
Other: Photodynamic therapy — A number of studies have reported that PDT can accelerate wound healing by inactivating local bacterial infection and colonization of bacterial biofilm, promoting wound re-epithelialization.
  Arms: Group 2 (Grp.2); Group 3 (Grp.3)
Other: Hydrogel dressing — Hydrogel dressing is widely applied in clinical practice to improve the regeneration ability of wound granulation tissue, promote the division and migration of epithelial cells, speed up wound healing and relieve the pain.
  Arms: Group 1 (Grp.1); Group 3 (Grp.3)

SUMMARY:
63 patients with chronic infectious wounds were enrolled in the controlled study. They were randomly divided into three groups equally. Group 1 (Grp.1): The patients received hydrogel dressing change at three days intervals. Group 2 (Grp.2): The patients received ALA-PDT treatment at ten days intervals for 4 sessions. Groups 3 (Grp.3): The patients received ALA-PDT at ten days intervals for 4 sessions combined with hydrogel dressing change every three days intervals. The wound healing rate, total effective rate, patient satisfaction, adverse reaction, and recurrence were assessed in all groups.

DETAILED DESCRIPTION:
Randomly divide the enrolled patients into three groups for treatment by utilizing SAS software (SAS Institute, Cary, NC, U.S.A.). Initially, the wound pus and secretions were washed three times with a sterile saline solution. Subsequently, surgical instruments were employed to debride the wound, particularly the necrotic tissue, as well as any carrion and foreign bodies within the wound bed and cavity, with care being taken to avoid injury to nerves and blood vessels in the surrounding area. Grp.1 was covered with hydrogel dressing (PAUL HARTMANN AG, Germany) and replaced 2-3 times a week with topical mupirocin ointment three times a day. Grp.2 received photodynamic therapy only. Grp.3 accepted PDT, then coated with hydrogel dressing as mentioned above. The treatment protocol of PDT is described as follows: after thorough debridement, ALA (Shanghai Fudan-Zhang jiang Bio-Pharmaceutical Co. Ltd, China) in an oil-in-water emulsion was smeared on the wound. After covering with dark plastic film for 3h, the wounds were illuminated by a light-emitting diode (LED) red light (Shenzhen Lifotronic Technology Co., Ltd, China). After the operation, a cold ice compress can be used to relieve the swelling and pain. Then, the hydrogel was uniformly applied to the wound and its surroundings (Grp.3). Grp.2 and Grp.3 received PDT at an interval of ten days for 4 sessions. In all groups, treatment responses and adverse reactions were recorded. All patients received the treatment as mentioned above and then evaluated the clinical outcome. After the end of the treatment, all patients returned for follow up at weeks 2, 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients with chronic wounds caused by trauma or surgery who failed to heal after traditional formal medical treatment at least over three months;
* 2) Patients with stable vital signs who had no systemic medical disease and did not take glucocorticoids, immunosuppressive agents, or anticoagulants during the entire treatment process;
* 3) Participants provided signed informed consent, were able to comply with the program, were willing to participate in follow-up, and were able to cooperate in the observation of adverse events and efficacy;
* 4) The diameter of the skin wound should not exceed 10 centimeters.

Exclusion Criteria:

* 1) Patients are allergic to ALA;
* 2) Women with recent fertility, pregnancy or lactation plans;
* 3) Patients with deepening wounds or worsening infections;
* 4) Poor compliance leading to an inability to complete the treatment in its entirety;
* 5) Cutaneous ulcer caused by vascular disease, autoimmune diseases, metabolic diseases, local or metastatic malignant tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate | Up to 12 weeks after the end of the treatment.
  Panoramic photographs of the wounds were taken by the same observer at each treatment and return visit using a digital camera, and the wound area was recorded using Image-Pro Plus 6.0 software. Wound size on the first day of treatment was considered to be 100%. The change in wound area size was compared to the initial before treatment and calculated as a percentage reduction.
The total effectiveness rate | Up to 12 weeks after the end of the treatment.
  The evaluation criteria were as follows: 1) If the wound area is completely healed, treatment was considered "significantly effective" (SE); 2) if the wound area was at least 50% healed, treatment was considered "effective" (E); 3) If the wound area was healed 30 - 50%, the treatment is considered as "improved" (IMP); 4) If the wound area is healed less than 30%, it is considered as "ineffective" (INE). "The total effectiveness rate" (Et) was calculated from the equation as follows:
  Et = (NSE+NE)/Nt × 100% NSE = the number of patients belonging to the SE groups NE = the number of patients belonging to the E groups Nt = the total number of patients
Patient satisfaction | Up to 12 weeks after the end of the treatment.
  Patients were surveyed about their level of satisfaction with the results after 12 weeks following the final course of treatment with the results as "satisfied," "somewhat satisfied," "somewhat dissatisfied," or "dissatisfied."

OTHER OUTCOMES:
Adverse effects | Up to 12 weeks after the end of the treatment.
  The severity (absent; mild; moderate; severe) and duration of adverse reactions such as pain, burning sensation, erythema, oedema and pigmentation, treatment measures and efficacy were meticulously documented at each treatment and follow-up.
Recurrence | Up to 12 weeks after the end of the treatment.
  Patients were surveyed about the recurrence after 12 weeks following the final course of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yin, MD, PhD, Principal Investigator — Southwest Hospital, Third Military Medical University, Chongqing, 400038, China
Locations (1):
- Department of Dermatology, Southwest Hospital, Third Military Medical University (Army Medical University), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nesi-Reis V, Lera-Nonose DSSL, Oyama J, Silva-Lalucci MPP, Demarchi IG, Aristides SMA, Teixeira JJV, Silveira TGV, Lonardoni MVC. Contribution of photodynamic therapy in wound healing: A systematic review. Photodiagnosis Photodyn Ther. 2018 Mar;21:294-305. doi: 10.1016/j.pdpdt.2017.12.015. Epub 2017 Dec 28. PMID 29289704
- [Background] Khorsandi K, Hosseinzadeh R, Esfahani H, Zandsalimi K, Shahidi FK, Abrahamse H. Accelerating skin regeneration and wound healing by controlled ROS from photodynamic treatment. Inflamm Regen. 2022 Oct 4;42(1):40. doi: 10.1186/s41232-022-00226-6. PMID 36192814
- [Background] Sies H, Jones DP. Reactive oxygen species (ROS) as pleiotropic physiological signalling agents. Nat Rev Mol Cell Biol. 2020 Jul;21(7):363-383. doi: 10.1038/s41580-020-0230-3. Epub 2020 Mar 30. PMID 32231263
- [Background] Morley S, Griffiths J, Philips G, Moseley H, O'Grady C, Mellish K, Lankester CL, Faris B, Young RJ, Brown SB, Rhodes LE. Phase IIa randomized, placebo-controlled study of antimicrobial photodynamic therapy in bacterially colonized, chronic leg ulcers and diabetic foot ulcers: a new approach to antimicrobial therapy. Br J Dermatol. 2013 Mar;168(3):617-24. doi: 10.1111/bjd.12098. Epub 2013 Jan 18. PMID 23066973
- [Background] Xu Y, Chen H, Fang Y, Wu J. Hydrogel Combined with Phototherapy in Wound Healing. Adv Healthc Mater. 2022 Aug;11(16):e2200494. doi: 10.1002/adhm.202200494. Epub 2022 Jul 6. PMID 35751637